CLINICAL TRIAL: NCT01718210
Title: GM-CSF Supplemented Medium for IVF Embryo Growth in Patients With Recurrent Implantation Failure
Brief Title: Use of GM-CSF Supplemented IVF Medium in Patients With Recurrent Implantation Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HC0005
Record Dates: First submitted 2012-03-02; First posted 2012-10-31 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Infertility
Keywords: GM-CSF; recurrent implantation failure; pregnancy rate; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GM-CSF medium (Experimental): patient's embryos are incubated after fertilization with mediun supplemented with GM-CSF
  Interventions: Drug: GM-CSF medium
- CONTROL (Placebo Comparator): 50 women with recurrent implantation failure (at leat three previous IVF attempts failed with at least 8 good embryos transferred in uterus)that the obtained with IVF are incubated with a standard medium for IVF, and utilized as control group.
  Interventions: Drug: CONTROL

INTERVENTIONS:
Drug: GM-CSF medium — incubation of IVF embryos with a specific medium containing GM-CSF
  Other Names: Embryogen
  Arms: GM-CSF medium
Drug: CONTROL — group of controls treated with a standard IVF medium
  Other Names: NORMAL MEDIUM
  Arms: CONTROL

SUMMARY:
The purpose of this study is to determine whether in Assisted Reproductive Technologies the use of culture medium supplemented with GM-CSF, a growth factor working on stem cells, may improve the embryo implantation in patients experiencing recurrent implantation failure in IVF cycles.

DETAILED DESCRIPTION:
In Assisted Reproductive Technologies the rate of pregnancy for cycle and the implantation rate remain low nevertheless the improvement in the last years. In particular there are a group of patients, in young reproductive age, experiencing recurrent implantation failure, nevertheless the good embryos produced and transferred. Recently, it has been showed that culture medium supplemented with GM-CSF, may improve the embryo outcomes in IVF. In this trial the investigators will test the potential benefits of this culture medium on embryos of patients experiencing recurrent implantation failure. 100 women with recurrent implantation failure, at least three failed previous IVF attempts with at least 8 good embryos transferred no more than 40 years old will be selected. These patients will be assigned to two arms, one experimental and one other of control by a computer generated sequence. After the oocyte retrieval and fertilization by ICSI procedure, the fertilised oocyte (2PN)will cultured with the GM-CSF supplemented culture medium (EmbryoGen, Origio, Denmark), or in normal culture in micro drop of 30microliters under oil until the day of transfer (day three or 8 cells sage embryos). A maximum of three embryos will be transferred. The pregnancy rate the implantation rate will be the outcomes considered

ELIGIBILITY:
Inclusion Criteria:

* woman age 40 years old or less,
* 3 or more consecutive previous failed IVF cycles with a total of at least 8 good embryos replaced in uterus

Exclusion Criteria:

* chromosomal defects in the couple,
* metabolic diseases (diabetes, etc),
* other genetic diseases (thalassemia, cystic fibrosis, etc.)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 9 months
  The number of patients become pregnant after IVF where GM-CSF medium is used, compared with the number of patients become pregnant in the control group

SECONDARY OUTCOMES:
Implantation rate | 9 months
  number of embryos implanted

CONTACTS AND LOCATIONS:
Overall Officials: Marco Sbracia, MD, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (1):
- Villa Salaria Fisiopatologia Riproduzione, Rome, Italy